CLINICAL TRIAL: NCT06321224
Title: Effects of Breathing Exercises on Women With Primary Dysmenorhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/03/08
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The exercise group will be given breathing exercises
  Interventions: Other: Breathing exercises
- Control group (Other): The control group will be asked to continue their routine lives.
  Interventions: Other: Control

INTERVENTIONS:
Other: Breathing exercises — Breathing exercises will be performed 3 days a week during 2 menstrual periods.
  Arms: Exercise group
Other: Control — No intervention will be made to the control group and they will be asked to continue their routine lives.
  Other Names: Routine live
  Arms: Control group

SUMMARY:
The aim of this study is to examine the effects of breathing exercises in women with primary dysmenorrhea.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is the most common gynecological disorder and constitutes a serious health and economic problem. PD is defined as painful menstrual cramps in the lower abdomen during or a few days before the menstrual period with no detectable organic disease. Breathing exercises are an effective method for pain relief. However, breathing exercises need to be examined in PD management.

ELIGIBILITY:
Inclusion Criteria:

* Having PD symptoms according to the Primary Dysmenorrhea Consensus criteria,
* Having menstrual pain intensity of 4 or higher according to the Visual Analog Scale in the last 6 months,
* Having a regular menstrual cycle (28±7 days)
* Volunteering to participate in the study.

Exclusion Criteria:

* Being pregnant or suspected of pregnancy,
* Using oral contraceptives or antidepressants in the last 6 months,
* Using intrauterine devices,
* Having a history of other gynecological diseases
* Having pulmonary, neurological and/or systemic disease,
* Having undergone abdominal or cardiothoracic surgery within the last year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Primary dysmenorrhea is a gynecological problem that can be seen in most women.
Enrollment: 42 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Menstrual pain intensity | After 2 menstrual periods
  Menstrual pain intensity will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0" = "no pain", while "10" = "unbearable pain".

SECONDARY OUTCOMES:
Menstrual symptoms | After 2 menstrual periods
  Menstrual symptoms will be measured with the Menstrual Symptom Questionnaire, consistng of 24 items.The total score is 120 points. An increase in the mean score indicates an increase in the severity of menstrual symptoms.
Life quality | After 2 menstrual periods
  Life quality will be evaluated with Dysmenorrhea Impact Scale. The 13-item structure of the scale is scored between 13-65 in total. As the scores obtained from the scale increase, the level of menstruation-related influence in people's lives increases
Stress level | After 2 menstrual periods
  Stress level will be evaluated with Perceived Stress Scale, consisting of a total of 14 items. The scale is scored between 0-56 in total. A high score from the scale indicates that the person has an increased perception of stress.
Sleep quality | After 2 menstrual periods
  Sleep quality will be evaluated with Pittsburgh Sleep Quality Index, consisting of 19 items. The total score of the scale ranges from 0 to 21, and a high total score indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University